CLINICAL TRIAL: NCT01434992
Title: Detection of Helicobacter Pylori Infection by Non-magnifying High Resolution Endoscopy is Possible Within the Gastric Corpus
Brief Title: Detection of Helicobacter Pylori Infection by High Resolution Endoscopy
Status: Completed | Type: Observational
Sponsor: Kyunghee University Medical Center (Other)
Responsible Party: Principal Investigator, Jun-Hyung Cho, Clinical and research fellow, Kyunghee University Medical Center
Other Study IDs: KHU-HP-2011
Record Dates: First submitted 2011-09-14; First posted 2011-09-15 (Estimated); Last update posted 2012-04-20 (Estimated); Status verified 2012-04

CONDITIONS: Helicobacter-associated Gastritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Gastric mucosa for detecting Helicobacter pylori
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- H. pylori gastritis

SUMMARY:
Although endoscopic findings of H. pylori have been reported in the literature, there is still some debate over whether H. pylori-related gastritis can be diagnosed via endoscopic features alone. Most studies concluded that it is not possible to diagnose H. pylori-related gastritis on the basis of endoscopic findings. However, the resolution power of endoscopy has greatly improved in recent years and the exact examination of gastric mucosa was possible.

DETAILED DESCRIPTION:
Our study aimed to achieve the following: (1) describe the H. pylori-related mucosal pattern in the gastric corpus using high-definition endoscopy; (2) evaluate the diagnostic accuracy for H. pylori detection; (3) find the optimal biopsy site for rapid urease test (RUT); (4) validate the inter- and intraobserver agreement in the assessment of endoscopic patterns.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent upper endoscopy

Exclusion Criteria:

* Age < 20 or > 70
* Severe systemic disease or advanced chronic liver disease
* Medication history of NSAID, PPI, H2 blockers or antibiotics
* History of H. pylori eradication therapy
* History of gastric surgery
* Recent history of upper GI bleeding
* Gastric or duodenal ulcer (including old scar change) during endoscopy
* Anemia (Hemoglobin level < 10mg/dL)
* Pangastritis

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent upper endoscopy in the Kyung Hee University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 585 (Actual)
Dates: Start 2011-08; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Diagnosis accuracy for predicting of Helicobacter pylori infection status | 1 day

SECONDARY OUTCOMES:
Assessment of the clinicopathologic factors related to correct diagnosis | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Jun-Hyung Cho, M.D., Principal Investigator — Kyung Hee University Hospital
Locations (1):
- Kyung Hee University Hospital, Seoul, South Korea

REFERENCES:
- [Background] Bah A, Saraga E, Armstrong D, Vouillamoz D, Dorta G, Duroux P, Weber B, Froehlich F, Blum AL, Schnegg JF. Endoscopic features of Helicobacter pylori-related gastritis. Endoscopy. 1995 Oct;27(8):593-6. doi: 10.1055/s-2007-1005764. PMID 8608753
- [Background] Redeen S, Petersson F, Jonsson KA, Borch K. Relationship of gastroscopic features to histological findings in gastritis and Helicobacter pylori infection in a general population sample. Endoscopy. 2003 Nov;35(11):946-50. doi: 10.1055/s-2003-43479. PMID 14606018
- [Background] Mihara M, Haruma K, Kamada T, Komoto K, Yoshihara M, Sumii K, Kajiyama G. The role of endoscopic findings for the diagnosis of Helicobacter pylori infection: evaluation in a country with high prevalence of atrophic gastritis. Helicobacter. 1999 Mar;4(1):40-8. doi: 10.1046/j.1523-5378.1999.09016.x. PMID 10352086
- [Derived] Cho JH, Chang YW, Jang JY, Shim JJ, Lee CK, Dong SH, Kim HJ, Kim BH, Lee TH, Cho JY. Close observation of gastric mucosal pattern by standard endoscopy can predict Helicobacter pylori infection status. J Gastroenterol Hepatol. 2013 Feb;28(2):279-84. doi: 10.1111/jgh.12046. PMID 23189930